CLINICAL TRIAL: NCT03421041
Title: A RCT Study of Value of Dexamethasone Used in Ovulation Induction
Brief Title: Study of Value of Dexamethasone Used in Ovulation Induction
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: protocol change
Sponsor: Reproductive & Genetic Hospital of CITIC-Xiangya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCYJ-201801
Record Dates: First submitted 2018-01-29; First posted 2018-02-05 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-01

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female | interventions — Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexamethasone group (Experimental)
  Interventions: Drug: Dexamethasone Oral Tablet
- control group (No Intervention)

INTERVENTIONS:
Drug: Dexamethasone Oral Tablet — Dexamethasone Oral Tablet，0.75mg/tablet
  Arms: Dexamethasone group

SUMMARY:
This study intends to solve the following problems: whether use dexamethasone can obviously decrease transplant cancelling probability in fresh embryo transplant cycle or not, reduce time and frequency going to hospital repeatedly for patients need frozen embryo transplant or not, and reduce the economic burden for patients or not; By comparing pregnancy rate of single transplant, hope to make clear in IVF-ET treatment for patients progesterone increases to a certain level whether it is a good choice to transfer fresh embryo after dexamethasone treatment, or frozen embryo transplant is better.

ELIGIBILITY:
Inclusion Criteria:

- female, 18 years old≤age≤35 years old, 18≤BMI≤25, standard patient, menstrual regularity

Exclusion Criteria:

Hyperprolactinemia, Thyroid dysfunction, uterine malformation ( inadequacy mediastinal uterus ≥1.0cm, Unicornate uterus, double uterus, T Angle of uterus, etc.), uterus adhesion, untreated hydrosalpinx , hysteromyoma（ hysteromyoma≥1.0 cm, and/or endometrial hysteromyoma≤1 cm), endometriosis, diabetes, hypertension, adrenal cortex hyperplasia, Cushing's syndrome, a pituitary amenorrhea

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
cumulative pregnancy rate per oocyte retrieval cycle | Until 28 day after embryo transferred
  cumulative pregnancy rate per oocyte retrieval cycle

CONTACTS AND LOCATIONS:
Locations (1):
- Reproductive & Genetic Hospital of CITIC-XIANGYA, Changsha, Hunan, China